CLINICAL TRIAL: NCT06214975
Title: The Effects of EXOPULSE Mollii Suit on Motor Functions in Patients With Stroke (EXOSTROKE 2)"
Brief Title: EXOPULSE Mollii Suit, Motor Function & Stroke (EXOSTROKE 2)
Acronym: EXOSTROKE2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheikh Shakhbout Medical City (Other)
Responsible Party: Principal Investigator, Naji Joseph Riachi, Principal Investigator, Sheikh Shakhbout Medical City
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EXOSTROKE2
Record Dates: First submitted 2023-11-20; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Stroke; Spasticity, Muscle; Spastic
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXOPULSE Mollii Suit Stimulation Active (Active Comparator): This will be the EXOPULSE Mollii Suit Active Stimulation. Stimulation will go on for 60 minutes while control unit is on for 60 minutes
  Interventions: Device: EXOPULSE Mollii Suit Stimulation
- EXOPULSE Mollii Suit Stimulation Sham (Sham Comparator): This will be the EXOPULSE Mollii Suit Sham Stimulation. Stimulation will go on for 1 minute then it turns off while the control unit will remain on for total of 60 minutes.
  Interventions: Device: EXOPULSE Mollii Suit Stimulation

INTERVENTIONS:
Device: EXOPULSE Mollii Suit Stimulation — We designed a randomized crossover, sham-controlled, double-blind trial to demonstrate the improvement of motor functions and stroke related symptoms following a single session of "active" versus "sham" EXOPULSE Mollii suit stimulation. in phase 1, the patient will receive two stimulations separated by a two-week washout period. The patients will be randomized to receive either active/sham or sham/active and both patients and investigators will be blinded to the order in which the stimulation will be given. A 2-week washout period should be enough to prevent a potential carry over effect. Two weeks after the end of phase 1, a second open label phase (phase 2) of this trial will be proposed to all patients where they will receive active stimulation every other day at home over four weeks (for a total of 14 sessions). This will help understand the long term effects of EXOPULSE Mollii suit stimulation on stroke related symptoms.

SUMMARY:
The goal of this clinical trial is to demonstrate the improvement of motor functions related symptoms in patients with stroke and spasticity using Exopulse Mollii suit stimulation.

The main questions it aims to answer are:

to evaluate the short-term impact of EXOPULSE Mollii suit on balance in adult patients with stroke and suffering from spasticity.

to assess the effects of Exopulse Mollii suit on spasticity, mobility, pain, fatigue and QoL.

.

Participants will participate in:

One baseline visit for inclusion during which the patient will undergo the first session (active or sham) along with evaluations (before and after the session) One visit after two weeks during which the patient will undergo the second session (active or sham) along with evaluations (before and after the session) One visit after two weeks of the second stimulation condition; the patients will undergo a third evaluation and receive the EXOPULSE Mollii Suit for the four-week open label phase and will use the suit at home for an active stimulation session every other day for four weeks.

One visit at the end of the open label phase to perform the fourth and last evaluation and return the EXOPULSE Mollii suit.

Researchers will compare both Active and Sham groups to demonstrate the improvement of motor functions related symptoms in patients with stroke and spasticity using Exopulse Mollii suit.

DETAILED DESCRIPTION:
The study is a randomized crossover, sham-controlled, double-blind trial to demonstrate the improvement of motor functions and stroke related symptoms following a single session of "active" versus "sham" EXOPULSE Mollii suit. A 2-week washout period should be enough to prevent a potential carry over effect. Two weeks after the end of this phase (phase 1), a second phase of this trial, an open label phase, will be proposed for all patients to understand the effects of EXOPULSE Mollii suit employed over 4 weeks (a session every other day for a total of 14 sessions) on stroke related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years.
* Having a clinical diagnosis of stroke since at least three months.
* Being able to walk freely or with the need of support (modified Rankin score ≤ 4).
* Able to understand verbal instructions.
* Having spasticity with a score of at least 1+ on the MAS.
* Having a BBS score ≤46 associated in the literature with a risk of fall.

Exclusion Criteria:

* Being included in another research protocol during the study period.
* Inability to undergo medical monitor for the study purposes due to geographical or social reasons.
* Having a cardiac stimulator, a ventriculoperitoneal shunt, an intrathecal baclofen pump or other contraindications to using EXOPULSE Mollii suit.
* Being pregnant.
* Having a change in their stroke pharmacological therapy in the last three months.
* Suffering from other somatic or neuropsychiatric diagnoses (e.g., arrhythmias, uncontrolled epilepsy, diseases causing osteoarticular and muscular pain).
* Having a body mass index above 35 Kg/m2.
* In case of the introduction of a medical device other than EXOPULSE Mollii suit during the study period.
* Patients under juridical protection.
* Prisoners.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Balance using Berg Balance Scale (BBS) | To be assessed at baseline.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in patients with stroke (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.
Balance using Berg Balance Scale (BBS) | To be assessed at week 2.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in patients with stroke (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.
Balance using Berg Balance Scale (BBS) | To be assessed at week 4.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in patients with stroke (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.
Balance using Berg Balance Scale (BBS) | To be assessed at week 8.
  Balance will be assessed using the 14-item Berg Balance Scale (BBS) which has good psychometric properties in patients with stroke (concurrent validity, interrater reliability). The scale rates the balance using 56 points, with higher scores indicating better balance abilities. A score equal to or below 45 is commonly associated with risk of fall across the literature.

SECONDARY OUTCOMES:
Visual Analog Score for spasticity. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Spasticity will be measured using a visual analog score from 0 to 10, 0 being no spasticity and 10 being the worst possible spasticity.
Visual Analog Score for pain. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Pain will be measured using a visual analog score from 0 to 10, 0 being no pain, to 10 being the worst possible pain.
EQ-5D-5L: EuroQol 5 Dimensions 5 Levels Quality of Life Questionnaire | Two weeks after the second stimulation and 4 weeks later at the end of phase 2.
Overall Clinical improvement | This to be assessed at baseline, then at week 2, and week 8.
  Evaluation of overall Clinical improvement will be done using the 7-point Clinical Global Impression (CGI). Patient will fill a questionnaire that will address their clinical situation as follows:
  Very much improved. Much improved. Slightly improved. No change. Slightly worse. Much worse. Very much worse.
  The score will range from 1-7, 1 being the best clinical outcome and 7 the worst.
Blinding Questionnaire | This to be assessed at baseline, then at week 2.
  Evaluation of patient's blinding to the type of stimulation in the crossover trial periods using a dedicated questionnaire. Patients will be asked whether they think they received the sham or active stimulation.
  No scale will be used for this measure.
Visual Analog Score for fatigue | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Fatigue will be measured using a visual analog score from 0 to 10, 0 being no fatigue, to 10 being the worst possible fatigue.
Muscle tone. | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Muscle tone will be evaluated by the Modified Ashworth Scale (MAS). Scores will range from 0 to 4, 0 being no increase or normal muscle tone, to 4 being rigidity in flexion or extension of muscles.
Fall Risk | Two weeks after the second stimulation and 4 weeks later at the end of phase 2.
  Fall risk will be assessed using the Falls Efficacy Scale-International scale. It is a 16-item scale, including a range of functional activities, that assesses the perceived risk of falling, using a score that will range from 1 to 4, 1 being not at all concerned to 4 being very concerned.
  Items are summed to a total score that will range from a minimum of 16 (no concern about falling) to a maximum of 64 (severe concern about falling).
Weight | Baseline.
  The patient weight will be measured and recorded in kilograms.
Height | Baseline
  The patient height will be measured and recorded in centimeters.
Time Up and Go (TUG) | This to be assessed at baseline, then at week 2, week 4 and week 8.
  Patients have to stand up from a chair when they hear the verbal instruction "go", walk a distance of 3 meters, turn around, walk back to the chair and sit down. Timing starts with the verbal instruction "go' and stops when the patients return to the seated position. The score consists of the time taken to complete the test activity, measured in seconds.
Body Mass Index (BMI) | Baseline
  The weight and height will be combined to report BMI in kg/m^2. BMI of 35 kg/m^2 or more will be used as an exclusion criterion for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Naji J Riachi, MD, Principal Investigator — SSMC
Locations (1):
- SSMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andringa A, van de Port I, van Wegen E, Ket J, Meskers C, Kwakkel G. Effectiveness of Botulinum Toxin Treatment for Upper Limb Spasticity Poststroke Over Different ICF Domains: A Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2019 Sep;100(9):1703-1725. doi: 10.1016/j.apmr.2019.01.016. Epub 2019 Feb 21. PMID 30796921
- [Background] Andersen IT, Harrison A, Broholm R, Harder A, Nielsen JB, Bulow J, Pingel J. Microvascularization is not a limiting factor for exercise in adults with cerebral palsy. J Appl Physiol (1985). 2018 Aug 1;125(2):536-544. doi: 10.1152/japplphysiol.00827.2017. Epub 2018 May 3. PMID 29722625
- [Background] Aree-uea B, Auvichayapat N, Janyacharoen T, Siritaratiwat W, Amatachaya A, Prasertnoo J, Tunkamnerdthai O, Thinkhamrop B, Jensen MP, Auvichayapat P. Reduction of spasticity in cerebral palsy by anodal transcranial direct current stimulation. J Med Assoc Thai. 2014 Sep;97(9):954-62. PMID 25536713
- [Background] Bakaniene I, Urbonaviciene G, Janaviciute K, Prasauskiene A. Effects of the Inerventions method on gross motor function in children with spastic cerebral palsy. Neurol Neurochir Pol. 2018 Sep-Oct;52(5):581-586. doi: 10.1016/j.pjnns.2018.07.003. Epub 2018 Jul 20. PMID 30061001
- [Background] Bar-On L, Molenaers G, Aertbelien E, Van Campenhout A, Feys H, Nuttin B, Desloovere K. Spasticity and its contribution to hypertonia in cerebral palsy. Biomed Res Int. 2015;2015:317047. doi: 10.1155/2015/317047. Epub 2015 Jan 11. PMID 25649546
- [Background] Barnes, M.P (2008). Upper Motor Neuone Syndrome and Spasticity: Clinical Management and Neurophysiology, Cambridge University Press, Cambridge, UK.
- [Background] Baude M, Nielsen JB, Gracies JM. The neurophysiology of deforming spastic paresis: A revised taxonomy. Ann Phys Rehabil Med. 2019 Nov;62(6):426-430. doi: 10.1016/j.rehab.2018.10.004. Epub 2018 Nov 28. PMID 30500361
- [Background] Bethoux F. Spasticity Management After Stroke. Phys Med Rehabil Clin N Am. 2015 Nov;26(4):625-39. doi: 10.1016/j.pmr.2015.07.003. Epub 2015 Sep 26. PMID 26522902
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Bonita R, Beaglehole R. Recovery of motor function after stroke. Stroke. 1988 Dec;19(12):1497-500. doi: 10.1161/01.str.19.12.1497. PMID 3201508
- [Background] Burke D, Wissel J, Donnan GA. Pathophysiology of spasticity in stroke. Neurology. 2013 Jan 15;80(3 Suppl 2):S20-6. doi: 10.1212/WNL.0b013e31827624a7. PMID 23319482
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Camak DJ. Addressing the burden of stroke caregivers: a literature review. J Clin Nurs. 2015 Sep;24(17-18):2376-82. doi: 10.1111/jocn.12884. Epub 2015 Jun 10. PMID 26095074
- [Background] Campbell WI, Lewis S. Visual analogue measurement of pain. Ulster Med J. 1990 Oct;59(2):149-54. PMID 2278111
- [Background] Cech, D. J., & Martin, S. T. (2012). Chapter 5 - Evaluation of Function, Activity, and Participation. In D. J. Cech & S. T. Martin (Eds.), Functional Movement Development Across the Life Span (Third Edition) (pp. 88-104). Saint Louis: W.B. Saunders.
- [Background] Chan PP, Si Tou JI, Tse MM, Ng SS. Reliability and Validity of the Timed Up and Go Test With a Motor Task in People With Chronic Stroke. Arch Phys Med Rehabil. 2017 Nov;98(11):2213-2220. doi: 10.1016/j.apmr.2017.03.008. Epub 2017 Apr 7. PMID 28392324
- [Background] Cogiamanian F, Ardolino G, Vergari M, Ferrucci R, Ciocca M, Scelzo E, Barbieri S, Priori A. Transcutaneous spinal direct current stimulation. Front Psychiatry. 2012 Jul 4;3:63. doi: 10.3389/fpsyt.2012.00063. eCollection 2012. PMID 22783208
- [Background] Denno MS, Gillard PJ, Graham GD, DiBonaventura MD, Goren A, Varon SF, Zorowitz R. Anxiety and depression associated with caregiver burden in caregivers of stroke survivors with spasticity. Arch Phys Med Rehabil. 2013 Sep;94(9):1731-6. doi: 10.1016/j.apmr.2013.03.014. Epub 2013 Mar 30. PMID 23548544
- [Background] Ertzgaard P, Alwin J, Sorbo A, Lindgren M, Sandsjo L. Evaluation of a self-administered transcutaneous electrical stimulation concept for the treatment of spasticity: a randomized placebo-controlled trial. Eur J Phys Rehabil Med. 2018 Aug;54(4):507-517. doi: 10.23736/S1973-9087.17.04791-8. Epub 2017 Oct 25. PMID 29072043
- [Background] Farid L, Jacobs D, Do Santos J, Simon O, Gracies JM, Hutin E. FeetMe(R) Monitor-connected insoles are a valid and reliable alternative for the evaluation of gait speed after stroke. Top Stroke Rehabil. 2021 Mar;28(2):127-134. doi: 10.1080/10749357.2020.1792717. Epub 2020 Jul 13. PMID 32654627
- [Background] Farrar JT, Troxel AB, Stott C, Duncombe P, Jensen MP. Validity, reliability, and clinical importance of change in a 0-10 numeric rating scale measure of spasticity: a post hoc analysis of a randomized, double-blind, placebo-controlled trial. Clin Ther. 2008 May;30(5):974-85. doi: 10.1016/j.clinthera.2008.05.011. PMID 18555944
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Flodstrom C, Viklund Axelsson SA, Nordstrom B. A pilot study of the impact of the electro-suit Mollii(R) on body functions, activity, and participation in children with cerebral palsy. Assist Technol. 2022 Jul 4;34(4):411-417. doi: 10.1080/10400435.2020.1837288. Epub 2021 Mar 29. PMID 33151822
- [Background] Gan SM, Tung LC, Tang YH, Wang CH. Psychometric properties of functional balance assessment in children with cerebral palsy. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):745-53. doi: 10.1177/1545968308316474. Epub 2008 Jul 21. PMID 18645187
- [Background] Ganapathy V, Graham GD, DiBonaventura MD, Gillard PJ, Goren A, Zorowitz RD. Caregiver burden, productivity loss, and indirect costs associated with caring for patients with poststroke spasticity. Clin Interv Aging. 2015 Nov 6;10:1793-802. doi: 10.2147/CIA.S91123. eCollection 2015. PMID 26609225
- [Background] Goldstein LB, Bertels C, Davis JN. Interrater reliability of the NIH stroke scale. Arch Neurol. 1989 Jun;46(6):660-2. doi: 10.1001/archneur.1989.00520420080026. PMID 2730378
- [Background] Golicki D, Niewada M, Buczek J, Karlinska A, Kobayashi A, Janssen MF, Pickard AS. Validity of EQ-5D-5L in stroke. Qual Life Res. 2015 Apr;24(4):845-50. doi: 10.1007/s11136-014-0834-1. Epub 2014 Oct 28. PMID 25347978
- [Background] Grassi B, Quaresima V. Near-infrared spectroscopy and skeletal muscle oxidative function in vivo in health and disease: a review from an exercise physiology perspective. J Biomed Opt. 2016 Sep;21(9):091313. doi: 10.1117/1.JBO.21.9.091313. PMID 27443955
- [Background] Gupta AD, Chu WH, Howell S, Chakraborty S, Koblar S, Visvanathan R, Cameron I, Wilson D. A systematic review: efficacy of botulinum toxin in walking and quality of life in post-stroke lower limb spasticity. Syst Rev. 2018 Jan 5;7(1):1. doi: 10.1186/s13643-017-0670-9. PMID 29304876
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Background] Johnson, M.I. (2008). Trancutaneous electrical nerve stimulation (TENS). In: Watson T, ed. Electrotherapy, Evidence based practice, 11th ed. Edinburgh:Churchill Livingstone, 253e296.
- [Background] Krause P, Edrich T, Straube A. Lumbar repetitive magnetic stimulation reduces spastic tone increase of the lower limbs. Spinal Cord. 2004 Feb;42(2):67-72. doi: 10.1038/sj.sc.3101564. PMID 14765138
- [Background] Kuo, C.-L., & Hu, G.-C. (2018). Post-stroke Spasticity: A Review of Epidemiology, Pathophysiology, and Treatments. Int J Gerontol. 12, 280-284.
- [Background] Lance, J. (1980). "Symposium synopsis," in Spasticity: Disordered Motor Control, R. G. Feldman, R. R. Young, and W. P. Koella, Eds., pp. 485-494, Yearbook Medical, Chicago, Ill, USA.
- [Background] Lecoffre C, de Peretti C, Gabet A, Grimaud O, Woimant F, Giroud M, Bejot Y, Olie V. National Trends in Patients Hospitalized for Stroke and Stroke Mortality in France, 2008 to 2014. Stroke. 2017 Nov;48(11):2939-2945. doi: 10.1161/STROKEAHA.117.017640. Epub 2017 Sep 29. PMID 28970279
- [Background] Lerdal A, Bakken LN, Kouwenhoven SE, Pedersen G, Kirkevold M, Finset A, Kim HS. Poststroke fatigue--a review. J Pain Symptom Manage. 2009 Dec;38(6):928-49. doi: 10.1016/j.jpainsymman.2009.04.028. PMID 19811888
- [Background] Little WJ. The classic: Hospital for the cure of deformities: course of lectures on the deformities of the human frame. 1843. Clin Orthop Relat Res. 2012 May;470(5):1252-6. doi: 10.1007/s11999-012-2302-y. PMID 22402809
- [Background] Maeda N, Urabe Y, Murakami M, Itotani K, Kato J. Discriminant analysis for predictor of falls in stroke patients by using the Berg Balance Scale. Singapore Med J. 2015 May;56(5):280-3. doi: 10.11622/smedj.2015033. PMID 25678051
- [Background] Mai J, Pedersen E. Mode of action of dantrolene sodium in spasticity. Acta Neurol Scand. 1979 Jun;59(6):309-16. doi: 10.1111/j.1600-0404.1979.tb02941.x. PMID 158280
- [Background] Malanga G, Reiter RD, Garay E. Update on tizanidine for muscle spasticity and emerging indications. Expert Opin Pharmacother. 2008 Aug;9(12):2209-15. doi: 10.1517/14656566.9.12.2209. PMID 18671474
- [Background] Markus, H. (2008). Stroke: causes and clinical features. Medicine, 36, 586-91.
- [Background] McDougall J, Chow E, Harris RL, Mills PB. Near-infrared spectroscopy as a quantitative spasticity assessment tool: A systematic review. J Neurol Sci. 2020 May 15;412:116729. doi: 10.1016/j.jns.2020.116729. Epub 2020 Feb 10. PMID 32120130
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119
- [Background] Mills PB, Dossa F. Transcutaneous Electrical Nerve Stimulation for Management of Limb Spasticity: A Systematic Review. Am J Phys Med Rehabil. 2016 Apr;95(4):309-18. doi: 10.1097/PHM.0000000000000437. PMID 26829077
- [Background] Mukherjee A, Chakravarty A. Spasticity mechanisms - for the clinician. Front Neurol. 2010 Dec 17;1:149. doi: 10.3389/fneur.2010.00149. eCollection 2010. PMID 21206767
- [Background] Ng SS, Hui-Chan CW. The timed up & go test: its reliability and association with lower-limb impairments and locomotor capacities in people with chronic stroke. Arch Phys Med Rehabil. 2005 Aug;86(8):1641-7. doi: 10.1016/j.apmr.2005.01.011. PMID 16084820
- [Background] Nielsen JB, Petersen NT, Crone C, Sinkjaer T. Stretch reflex regulation in healthy subjects and patients with spasticity. Neuromodulation. 2005 Jan;8(1):49-57. doi: 10.1111/j.1094-7159.2005.05220.x. PMID 22151383
- [Background] Nordstrom B, Prellwitz M. A pilot study of children and parents experiences of the use of a new assistive device, the electro suit Mollii. Assist Technol. 2021 Sep 3;33(5):238-245. doi: 10.1080/10400435.2019.1579267. Epub 2019 Apr 4. PMID 30945989
- [Background] Palisano RJ, Cameron D, Rosenbaum PL, Walter SD, Russell D. Stability of the gross motor function classification system. Dev Med Child Neurol. 2006 Jun;48(6):424-8. doi: 10.1017/S0012162206000934. PMID 16700931
- [Background] Palmcrantz S, Pennati GV, Bergling H, Borg J. Feasibility and potential effects of using the electro-dress Mollii on spasticity and functioning in chronic stroke. J Neuroeng Rehabil. 2020 Aug 10;17(1):109. doi: 10.1186/s12984-020-00740-z. PMID 32778118
- [Background] Pandyan AD, Gregoric M, Barnes MP, Wood D, Van Wijck F, Burridge J, Hermens H, Johnson GR. Spasticity: clinical perceptions, neurological realities and meaningful measurement. Disabil Rehabil. 2005 Jan 7-21;27(1-2):2-6. doi: 10.1080/09638280400014576. No abstract available. PMID 15799140
- [Background] Perrot A, Castanier C, Maillot P, Zitari H. French validation of the modified-falls efficacy scale (M-FES Fr). Arch Gerontol Geriatr. 2018 Sep-Oct;78:233-239. doi: 10.1016/j.archger.2018.07.001. Epub 2018 Jul 4. PMID 30025268
- [Background] Picelli A, Santamato A, Chemello E, Cinone N, Cisari C, Gandolfi M, Ranieri M, Smania N, Baricich A. Adjuvant treatments associated with botulinum toxin injection for managing spasticity: An overview of the literature. Ann Phys Rehabil Med. 2019 Jul;62(4):291-296. doi: 10.1016/j.rehab.2018.08.004. Epub 2018 Sep 13. PMID 30219307
- [Background] Rabchevsky AG, Kitzman PH. Latest approaches for the treatment of spasticity and autonomic dysreflexia in chronic spinal cord injury. Neurotherapeutics. 2011 Apr;8(2):274-82. doi: 10.1007/s13311-011-0025-5. PMID 21384222
- [Background] Ro T, Ota T, Saito T, Oikawa O. Spasticity and Range of Motion Over Time in Stroke Patients Who Received Multiple-Dose Botulinum Toxin Therapy. J Stroke Cerebrovasc Dis. 2020 Jan;29(1):104481. doi: 10.1016/j.jstrokecerebrovasdis.2019.104481. Epub 2019 Nov 4. PMID 31699575
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Stevenson T. Berg balance test. Phys Ther. 1996 Oct;76(10):1124, 1126. doi: 10.1093/ptj/76.10.1124. No abstract available. PMID 8863765
- [Background] Stinear C, Ackerley S, Byblow W. Rehabilitation is initiated early after stroke, but most motor rehabilitation trials are not: a systematic review. Stroke. 2013 Jul;44(7):2039-45. doi: 10.1161/STROKEAHA.113.000968. Epub 2013 May 28. No abstract available. PMID 23715959
- [Background] Roche N, Lackmy A, Achache V, Bussel B, Katz R. Effects of anodal transcranial direct current stimulation over the leg motor area on lumbar spinal network excitability in healthy subjects. J Physiol. 2011 Jun 1;589(Pt 11):2813-26. doi: 10.1113/jphysiol.2011.205161. Epub 2011 Apr 18. PMID 21502292
- [Background] Sommerfeld DK, Gripenstedt U, Welmer AK. Spasticity after stroke: an overview of prevalence, test instruments, and treatments. Am J Phys Med Rehabil. 2012 Sep;91(9):814-20. doi: 10.1097/PHM.0b013e31825f13a3. PMID 22760104
- [Background] Tuppin P, Riviere S, Rigault A, Tala S, Drouin J, Pestel L, Denis P, Gastaldi-Menager C, Gissot C, Juilliere Y, Fagot-Campagna A. Prevalence and economic burden of cardiovascular diseases in France in 2013 according to the national health insurance scheme database. Arch Cardiovasc Dis. 2016 Jun-Jul;109(6-7):399-411. doi: 10.1016/j.acvd.2016.01.011. Epub 2016 Apr 11. PMID 27079468
- [Background] Vivancos-Matellano F, Pascual-Pascual SI, Nardi-Vilardaga J, Miquel-Rodriguez F, de Miguel-Leon I, Martinez-Garre MC, Martinez-Caballero I, Lanzas-Melendo G, Garreta-Figuera R, Garcia-Ruiz PJ, Garcia-Bach M, Garcia-Aymerich V, Bori-Fortuny I, Aguilar-Barbera M; Spanish Group on Spasticity. [Guide to the comprehensive treatment of spasticity]. Rev Neurol. 2007 Sep 16-30;45(6):365-75. Spanish. PMID 17899519
- [Background] Wade DT. Measuring arm impairment and disability after stroke. Int Disabil Stud. 1989 Apr-Jun;11(2):89-92. doi: 10.3109/03790798909166398. PMID 2698395
- [Background] Ward AB. A literature review of the pathophysiology and onset of post-stroke spasticity. Eur J Neurol. 2012 Jan;19(1):21-7. doi: 10.1111/j.1468-1331.2011.03448.x. Epub 2011 Jun 27. PMID 21707868
- [Background] WHO (2004). The atlas of heart disease and stroke / Judith Mackay and George Mensah ; with Shanthi Mendis and Kurt Greenland. World Health Organization. https://apps.who.int/iris/handle/10665/43007
- [Background] WHO (2019). Accident vasculaire cérébral (AVC). Disponible sur http://www.who.int/topics/cerebrovascular_accident/fr/
- [Background] Winkler T, Hering P, Straube A. Spinal DC stimulation in humans modulates post-activation depression of the H-reflex depending on current polarity. Clin Neurophysiol. 2010 Jun;121(6):957-61. doi: 10.1016/j.clinph.2010.01.014. Epub 2010 Feb 11. PMID 20153248
- [Background] Wu D, Qian L, Zorowitz RD, Zhang L, Qu Y, Yuan Y. Effects on decreasing upper-limb poststroke muscle tone using transcranial direct current stimulation: a randomized sham-controlled study. Arch Phys Med Rehabil. 2013 Jan;94(1):1-8. doi: 10.1016/j.apmr.2012.07.022. Epub 2012 Aug 7. PMID 22878231
- [Background] Zawawi NSM, Aziz NA, Fisher R, Ahmad K, Walker MF. The Unmet Needs of Stroke Survivors and Stroke Caregivers: A Systematic Narrative Review. J Stroke Cerebrovasc Dis. 2020 Aug;29(8):104875. doi: 10.1016/j.jstrokecerebrovasdis.2020.104875. Epub 2020 May 23. PMID 32689648
- [Background] Zorowitz RD, Gillard PJ, Brainin M. Poststroke spasticity: sequelae and burden on stroke survivors and caregivers. Neurology. 2013 Jan 15;80(3 Suppl 2):S45-52. doi: 10.1212/WNL.0b013e3182764c86. PMID 23319485